CLINICAL TRIAL: NCT04876248
Title: Phase 2 Trial of Belantamab Mafodotin Consolidation Treatment in Patients With Multiple Myeloma and MRD Positivity After Autologous Stem Cell Transplantation
Brief Title: Belantamab Mafodotin and Lenalidomide for the Treatment of Multiple Myeloma in Patients With Minimal Residual Disease Positive After Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 797720; NCI-2021-02349 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 797720 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (belantamab mafodotin, lenalidomide) (Experimental): Patients receive belantamab mafodotin IV over 30 minutes on day 1 and lenalidomide PO QD on days 1-28. Treatment repeats every 8 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Belantamab Mafodotin; Drug: Lenalidomide

INTERVENTIONS:
Biological: Belantamab Mafodotin — Given IV
  Other Names: Belantamab Mafodotin-blmf; Blenrep; GSK2857916; J6M0-mcMMAF
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial investigates the effect of belantamab mafodotin and lenalidomide on minimal residual disease negative rates in patients with multiple myeloma with minimal residual disease positive after stem cell transplant. Belantamab mafodotin is a monoclonal antibody, called belantamab, linked to a chemotherapy drug, called mafodotin. Belantamab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as B-cell maturation antigen (BCMA) receptors, and delivers mafodotin to kill them. Lenalidomide may help block the formation of growths that may become cancer, and is used as a standard of care treatment for multiple myeloma. Giving belantamab mafodotin and lenalidomide may help to maintain minimal residual disease negativity in patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the minimal residual disease (MRD) negative rate after 6 cycles of post autologous stem cell transplant consolidation with belantamab mafodotin and lenalidomide.

SECONDARY OBJECTIVE:

I. Assess sustained MRD negative rate, progression free survival (PFS) and overall survival (OS).

OUTLINE:

Patients receive belantamab mafodotin intravenously (IV) over 30 minutes on day 1 and lenalidomide orally (PO) once daily (QD) on days 1-28. Treatment repeats every 8 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 12 weeks and the periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age at time of consent
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically or cytologically confirmed diagnosis of multiple myeloma (MM) as defined according to International Myeloma Working Group (IMWG), 2016 criteria, and

  * Patient is considered transplant eligible, and
  * Is not MRD negative complete response (CR) after high dose chemotherapy
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L (within 14 days of first dose of study treatment)
* Hemoglobin >= 8.0 g/dL (within 14 days of first dose of study treatment)
* Platelets >= 75 X 10^9/L (within 14 days of first dose of study treatment)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (isolated bilirubin >= 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) (within 14 days of first dose of study treatment)
* Alanine aminotransferase (ALT) =< 2.5 X ULN or < 5 times ULN if documented liver infiltration (within 14 days of first dose of study treatment)
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/ 1.73 m^2 (within 14 days of first dose of study treatment)
* Spot urine (albumin/creatinine ratios (spot urine) < 500 mg/g (56 mg/mmol) OR urine dipstick Negative/trace (if >= 1+ only eligible if confirmed =< 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void) (within 14 days of first dose of study treatment)
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period
* Female participants of childbearing potential are to have a negative serum pregnancy test within 24 hours before the first dose of study intervention
* A male participant must agree to use an adequate method of contraception (as described below) during the treatment period and for at least 6 months after the last dose of study treatment to allow for clearance of any altered sperm, along with the following:

  * Refrain from donating sperm PLUS either:

    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
    * Must agree to use contraception/barrier
* All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be =< grade 1 at the time of enrolment except for alopecia
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Evidence of active bleeding requiring intervention within the last four weeks prior to first dose of study treatment
* Current corneal epithelial disease except mild changes in corneal epithelium
* Any major surgery within the last four weeks of first dose of study treatment
* Use of contact lenses while participating in this study
* Participant must not have had plasmapheresis within 7 days prior to first dose of study treatment
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect patient's safety). Patients with isolated proteinuria resulting from MM are eligible
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with patient's safety or compliance to the study procedures
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if patient otherwise meets entry criteria
* Malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction
* Evidence of cardiovascular risk including any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant electrocardiography (EKG) abnormalities such as 2nd degree (type II) or 3rd degree atrioventricular (AV) block.
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within two months of first dose.
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system.
  * Uncontrolled hypertension
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin or lenalidomide
* Active infection requiring antibiotic, antiviral, or antifungal treatment
* Known human immunodeficiency virus (HIV) infection
* Presence of hepatitis B surface antigen (HBsAg), at or within 3 months of registration Note: If Hepatitis B core antibody (HBcAb) present, see additional monitoring recommendations
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at or within 3 months prior registration. Note: Patients with positive hepatitis C antibody due to prior resolved disease can be eligible, only if a confirmatory negative hepatitis C RNA test is obtained.

  * Note: Hepatitis RNA testing is optional and patients with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing
* Best corrected visual acuity in the worst seeing eye worse than 20/100 (Snellen equivalent). Participants with vision worse than 20/100 due to a treatable condition (e.g., cataract) may be considered on an individual case basis within 6 months before registration
* Use of an investigational drug within 14 days of first dose of study treatment or five half-lives, whichever is shorter, preceding the first dose of study drug. Prior treatment with a monoclonal antibody within 30 days of first dose of study treatment
* Previously progressed on treatment with belantamab mafodotin
* Pregnant or lactating female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negative rate | After 6 cycles of post-transplant consolidation with belantamab mafodotin and lenalidomide (1 cycle = 8 weeks)
  A 90% confidence interval about true 6-month post-consolidation MRD negative rate will be obtained.

SECONDARY OUTCOMES:
Sustained MRD negative rate | At 1 year after end of consolidation
Progression-free survival | Time from the start of consolidation therapy until disease progression death, due to disease, or last disease evaluation, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, with estimates of the median obtained with 90% confidence intervals.
Overall survival | Time from the start of consolidation until death due to any cause or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods, with estimates of the median obtained with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Mohan M, Gundarlapalli S, Szabo A, Yarlagadda N, Kakadia S, Konda M, Jillella A, Fnu A, Ogunsesan Y, Yarlagadda L, Thalambedu N, Munawar H, Graziutti M, Al Hadidi S, Alapat D, Thanendrarajan S, Zangari M, van Rhee F, Schinke C. Tandem autologous stem cell transplantation in patients with persistent bone marrow minimal residual disease after first transplantation in multiple myeloma. Am J Hematol. 2022 Jun 1;97(6):E195-E198. doi: 10.1002/ajh.26530. Epub 2022 Mar 21. No abstract available. PMID 35285981
- [Derived] Mohan M, Hari P, Szabo A, Dhakal B, Chhabra S, D'Souza A. Long term follow up of newly diagnosed multiple myeloma patients treated with pembrolizumab consolidation post-autologous stem cell transplantation. Leuk Res. 2021 Oct;109:106648. doi: 10.1016/j.leukres.2021.106648. Epub 2021 Jun 23. No abstract available. PMID 34182226